CLINICAL TRIAL: NCT01846988
Title: Efficacy of Auto-adjustable Positive Airway Pressure (APAP) in Pediatric Patients With Obstructive Sleep Apnea (OSA).
Brief Title: Comparing Auto-adjustable Positive Airway Pressure to Continuous Positive Airway Pressure in Children With Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CIN001APAP
Record Dates: First submitted 2013-04-22; First posted 2013-05-06 (Estimated); Results first posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Pediatric Obstructive Sleep Apnea; Auto PAP; Auto-adjustable Positive Airway Pressure; APAP; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 crossover treatment (Active Comparator): crossover treatment (REMstar Auto A-Flex) Placed on REMstar Auto A-Flex machine with APAP settings for 4-8 weeks then randomized to 4 weeks APAP settings then 4 weeks CPAP settings.
  Interventions: Device: crossover treatment (REMstar Auto A-Flex)
- Group 2 crossover treatment (Active Comparator): crossover treatment (REMstar Auto A-Flex) Placed on REMstar Auto A-Flex machine with APAP settings for 4-8 weeks then randomized to 4 weeks CPAP settings then 4 weeks APAP settings.
  Interventions: Device: crossover treatment (REMstar Auto A-Flex)
- APAP pressurized comparison (Active Comparator): randomization periods for 6-8 weeks. An in-hospital APAP titration study will average 90th pressure percentile and average CPAP pressure derived from the device will be compared to the CPAP pressure determined by CPAP titration PSG. Subjects will then be randomized to Group 1 first, or Group 2 first, then crossover to the other group.
  Interventions: Device: crossover treatment (REMstar Auto A-Flex)

INTERVENTIONS:
Device: crossover treatment (REMstar Auto A-Flex) — All subjects will use same device with 4 week crossover of settings of APAP and CPAP
  Other Names: REMstar Auto A-Flex

SUMMARY:
The purpose of this research study is to determine if auto-adjustable positive airway pressure (APAP) is an effective way to treat obstructive sleep apnea (OSA) in children. APAP is a device similar to continuous positive airway pressure (CPAP) that delivers pressure to the upper airway (nose and throat) to keep the airway from collapsing while during sleep. The difference is that APAP adjusts the pressure throughout the night with changes in resistance during breathing, and CPAP gives the same amount of pressure the whole time it is worn. APAP is currently widely used to treat adults with OSA, however, this device has not yet been extensively studied in children.

There are two parts to this research study. Subjects will begin using APAP at the time of enrollment for 4 to 8 weeks. The investigators will compare the pressure measured by the APAP device over the 4-8 weeks with the pressure determined by a CPAP titration study. The titration study is a second overnight sleep study that is routinely ordered when a child with sleep apnea starts treatment with CPAP. It tells the doctor what CPAP setting should be used.

In the second part of this study The investigators will compare the effects of APAP with CPAP to see what is reported as more comfortable and is used during more hours of sleep. This part of the study will last about 8 weeks and each subject will use both CPAP and APAP for 4 weeks each.

Currently when someone is diagnosed with OSA there is a delay in starting treatment with CPAP until the results of the titration study are available. In this research, patients could be allowed to immediately start treatment with APAP. If APAP is found to be as safe and effective as regular CPAP, treatment with APAP could be used as an alternative to CPAP.

DETAILED DESCRIPTION:
This is a small clinical trial to test the feasibility of using APAP in children with sleep apnea.

Continuous positive airway pressure (CPAP) is commonly used to treat OSA by delivering a predetermined amount of positive pressure to the patient's upper airway in order to reduce the collapsibility of airway structures during sleep. The commonly accepted method for determining the appropriate pressure setting for children with OSA is through an in-hospital overnight CPAP titration study. Another commonly used treatment modality in adults with OSA is auto-adjustable positive airway pressure (APAP), in which airway patency is maintained by adjusting pressure delivery through the night depending on the needs of the patient as determined by the device. Benefits of APAP compared with CPAP include the ability to initiate therapy without an inpatient CPAP titration study, resulting in more prompt establishment of treatment and cost-savings. Patient adherence may also be significantly improved as the pressure delivered is appropriate for sleep stage and patient position, resulting in greater patient comfort. Utility and efficacy of APAP compared to CPAP have never been evaluated in the pediatric population.

The aim of this study is to establish APAP as an effective means of assessing CPAP pressure for OSA in children, and to determine if APAP therapy confers better treatment adherence and quality of life compared to traditional CPAP. The investigators hypothesize that APAP can effectively approximate the pressure determined by CPAP titration study, that APAP is superior to fixed CPAP in terms of treatment success, and that adherence to therapy will be improved with APAP compared to CPAP.

Forty patients aged 5-20 years will be enrolled in the study. These subjects will be recruited from the pediatric pulmonary or pediatric sleep clinic at Cincinnati Children's Hospital. Patients who are suspected of having OSA will be referred in the usual manner to the sleep center for diagnostic sleep study (PSG). Following the establishment of OSA diagnosis and subsequent enrollment in the study, the subject will begin therapy with APAP which will continue for 4 to 8 weeks. In that period of time the clinically ordered in-hospital CPAP titration study will be completed. The subject will then be randomized to either traditional fixed pressure CPAP at the pressure determined by in-hospital titration or APAP. The subject will receive 4 weeks of treatment in the randomized group (CPAP or APAP) then crossover to 4 weeks in the alternate group (CPAP or APAP). Both patient and researcher will be blinded to the randomization of pressure modality. The total study period will range from 12-16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 5 to 20 years of age
* apnea hypopnea index (AHI) of ≥5 or obstructive hypoventilation

Exclusion Criteria:

* significant cranio-facial abnormalities
* chromosomal abnormalities that would affect compliance
* cerebral palsy
* significant neurological disease or neuromuscular disease

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Narong Simakajornboon, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Neepa Gurbani, DO, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data at this time.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 15 subjects started study procedures. 5 subjects withdrew after completing the APAP pressurized comparison phase and only 10 subjects were randomized to crossover treatment. All randomized subjects completed the study. Data analysis includes the 5 withdrawals completing APAP pressurized comparison plus the 10 subjects completing study procedures.
Groups:
- APAP Pressurized Comparison: An in-hospital titration study will average 90th pressure percentile and average CPAP pressure derived from the device will be compared to the CPAP pressure determined by CPAP titration PSG. Subjects will then be randomized to Group 1 first, or Group 2 first, then crossover to the other group.
- Group 1: Randomized to APAP for 4 weeks followed by crossover to CPAP for 4 weeks after APAP settings for 4-8 weeks.
- Group 2: Randomized to CPAP for 4 weeks followed by crossover to APAP for 4 weeks after APAP settings for 4-8 weeks.
Period: APAP Pressurize Comparison (4-8 Weeks)
Arm/Group | APAP Pressurized Comparison | Group 1 | Group 2
Started | 15 | 0 | 0
Completed | 15 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Intervention #1 - 4 Weeks
Arm/Group | APAP Pressurized Comparison | Group 1 | Group 2
Started | 0 | 5 (Only 10 of 15 participants completing Comparison period started periods 1 & 2) | 5
Completed | 0 | 5 | 5
Not Completed | 0 | 0 | 0
Period: Intervention #2 - 4 Weeks
Arm/Group | APAP Pressurized Comparison | Group 1 | Group 2
Started | 0 | 5 | 5
Completed | 0 | 5 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data for all 15 subjects at baseline was analyzed.
Groups:
- APAP Pressurized Comparison: Comparison usage to determine APAP average 90% pressure (APAP P90) for initial treatment period and to assess adherence for randomization periods for 6-8 weeks or 4-6 weeks.
  Subjects will then be randomized to Group 1 first, or Group 2 first, then crossover to the other group.
- Group 1 Crossover Treatment: Randomized to APAP for 4 weeks followed by crossover to CPAP for 4 weeks after APAP settings for 4-8 weeks.
- Group 2 Crossover Treatment: Randomized to CPAP for 4 weeks followed by crossover to APAP for 4 weeks after APAP settings for 4-8 weeks.
- Total: Total of all reporting groups
Arm/Group | APAP Pressurized Comparison | Group 1 Crossover Treatment | Group 2 Crossover Treatment | Total
Number analyzed (Participants) | 15 | 0 | 0 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 0 | 0 | 15
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.3 (3.1) |  |  | 14.3 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 |  |  | 7
  Male | 8 |  |  | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15 |  |  | 15

OUTCOME MEASURES:

1. Primary Outcome: Difference Between Optimal Pressure (cm H2O) Derived From APAP run-in Period Versus Result of CPAP Titration Study
Description: The aim of this study is to establish APAP as an effective treatment modality for OSAS in the pediatric population. We hypothesize that APAP can effectively approximate the pressure determined by PSG CPAP titration as measured by the average 90th pressure percentile and average CPAP pressure delivered to the patient. The in-lab CPAP titration PSG following initial diagnosis of OSA is the current standard of therapy. APAP would potentially bridge the gap between the time of diagnosis and the follow up PSG for CPAP titration, allowing for more prompt intervention.
Time Frame: First visit after APAP run-in at 6-8 weeks
Population: The APAP pressure comparison group included 15 participants. After this initial period, 5 participants withdrew from the study. The remaining 10 participants were randomized to Group 1 or 2.
Measure: Mean (Standard Deviation); unit: cmH2O
Groups:
- APAP Pressure Comparison: APAP pressure comparison period was 6-8 weeks. APAP average 90th pressure percentile derived from machine download was compared to CPAP pressure determined by CPAP titration PSG. Subjects will then be randomized to Group 1 first, or Group 2 first, then crossover to the other group.
Arm/Group | APAP Pressure Comparison
Number analyzed (Participants) | 15
cmH2O
  APAP 90 percent pressure | 7.3 (2.6)
  CPAP titration PSG pressure | 9.4 (2.6)

2. Primary Outcome: Adherence Comparison of APAP vs.CPAP (% Days Device Used and % Days Device Used >4 Hours)
Description: Randomized crossover period comparison of adherence between APAP and CPAP calculated from therapy usage hours.
Time Frame: end of study visit at 12-16 weeks
Population: For data analysis we combined APAP data together and CPAP data together regardless of the order of randomization, yielding 10 subjects for APAP adherence and 10 subjects for CPAP adherence. In the data analysis below the column labeled Group 1 contains all APAP data and Group 2 contains all CPAP data.
Measure: Mean (Standard Deviation); unit: percentage of days
Groups:
- Group 1: Combined APAP data regardless of the order of randomization
- Group 2: Combined CPAP data regardless of order of randomization
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 10 | 10
percentage of days
  % days device used | 62.5 (27.2) | 61.4 (25.6)
  % days device used >4h | 42.7 (29.0) | 44.3 (29.4)

3. Secondary Outcome: Michigan Pediatric Sleep Questionnaire
Description: Comparison of Michigan pediatric sleep questionnaire score between baseline (at time of enrollment in the study) and each group (APAP, CPAP) after randomization period for the 10 subjects who completed the study. The scale range is from 0 to 1, Normal <0.33, at risk is 0.33-0.55 and >0.55 abnormal.
Time Frame: 12-16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: Michigan pediatric questionnaire score obtained at baseline at the time of enrollment into the study for subjects who were then randomized to APAP and CPAP.
- Group 1: Michigan pediatric sleep questionnaire score administered after APAP randomization period regardless of the order of randomization.
- Group 2: Michigan pediatric sleep questionnaire score administered after CPAP randomization period regardless of the order of randomization.
Arm/Group | Baseline | Group 1 | Group 2
Number analyzed (Participants) | 10 | 10 | 10
score on a scale | 0.65 (0.2) | 0.44 (0.2) | 0.39 (0.2)

4. Secondary Outcome: Epworth Sleepiness Scale Questionnaire
Description: Comparison of Epworth Sleepiness scale questionnaire score between baseline (at time of enrollment in the study) and each group (APAP, CPAP) after randomization period for the 10 subjects who completed the study. The scale range is from 0 to 24, with a value of 10 or greater suggesting significance for sleep disordered breathing.
Time Frame: 12-16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: Epworth sleepiness scale questionnaire data obtained at baseline at the time of enrollment into the study for subjects who were then randomized to APAP and CPAP.
- Group 1: Epworth sleepiness scale questionnaire data administered after APAP randomization period regardless of the order of randomization.
- Group 2: Epworth sleepiness scale questionnaire data administered after CPAP randomization period regardless of the order of randomization.
Arm/Group | Baseline | Group 1 | Group 2
Number analyzed (Participants) | 10 | 10 | 10
score on a scale | 10.3 (6.2) | 7.6 (5.0) | 7.2 (4.3)

5. Secondary Outcome: Comparison of Pediatric Quality of Life Inventory Questionnaire Score Between Baseline and Each Randomization Period
Description: Comparison of Pediatric Quality of Life Inventory questionnaire score between baseline (at time of enrollment in the study) and each group (APAP, CPAP) after randomization period for the 10 subjects who completed the study. The scale scores range between 0-100. Higher scores indicate better health related quality of life. Healthy: 81.34-100, at risk: 81.33-65.4, unhealthy <65.4
Time Frame: 12-16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: Pediatric Quality of Life Inventory questionnaire data obtained at baseline at the time of enrollment into the study for subjects who were then randomized to APAP and CPAP.
- Group 1: Pediatric Quality of Life Inventory questionnaire data administered after APAP randomization period regardless of the order of randomization.
- Group 2: Pediatric Quality of Life Inventory questionnaire data administered after CPAP randomization period regardless of the order of randomization.
Arm/Group | Baseline | Group 1 | Group 2
Number analyzed (Participants) | 10 | 10 | 10
score on a scale | 61.7 (17.9) | 65.9 (20.2) | 68.5 (18.3)

ADVERSE EVENTS:
Time Frame: From enrollment start until study completion, an average of 16 weeks
Description: The arms/groups are combined to maintain the format used for reporting outcomes. There were no adverse events to report in the study.
Arm/Group | APAP Pressurized Comparison | Group 1 Crossover Treatment | Group 2 Crossover Treatment
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/15 | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
Small sample size, small number of pre-adolescent subjects, and short term study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT01846988/Prot_SAP_000.pdf